CLINICAL TRIAL: NCT06916624
Title: Multicenter Study of 18F-Labeled NY104 for PET/CT Imaging in Renal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Qianfoshan Hospital (Other); Weifang People's Hospital (Other); Zibo Central Hospital (Other Government); Jining Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: QDFY-NM-25003
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Carcinoma (RCC); Clear Cell Renal Cell Carcinoma (ccRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-NY104 PET/CT scan
  Interventions: Radiation: 18F-NY104 PET/CT

INTERVENTIONS:
Radiation: 18F-NY104 PET/CT — The radionuclide ¹⁸F will serve as the tracer in this study. NY104 will be labeled with [¹⁸F]AlF to form the ¹⁸F-NY104 injection for use in this research.All participants will undergo ¹⁸F-NY104 PET scan.

SUMMARY:
Study on the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of 18F-NY104 PET/CT in diagnosing primary, recurrent, and metastatic lesions of renal cell carcinoma; and investigate the effect of oral low-dose CAIX inhibitor (Acetazolamide) on the tissue distribution of 18F-NY104 in renal cell carcinoma patients, particularly in the stomach and kidneys.

DETAILED DESCRIPTION:
Currently, the global population with kidney diseases exceeds 500 million, and the number of kidney disease patients in China is approximately 120 million, accounting for about 10.8% of the adult population. Among various kidney diseases, renal cell carcinoma (RCC) is the most severe kidney-destructive lesion. In recent years, the incidence of RCC in China has been increasing at an annual rate of approximately 3%, making it one of the most common malignant tumors in the urinary system. The disease is more prevalent in urban areas than rural regions, more frequent in males than females (gender ratio), with the high-risk age group being 45-65 years old. RCC is a highly aggressive tumor; about one-third of patients already present with metastasis at diagnosis, and over 40% of patients ultimately succumb to the disease. Currently, the etiology of RCC remains unclear. Early-stage RCC is asymptomatic but can be detected through health screenings. Compared to other cancers, RCC has a relatively better prognosis, yet 20%-40% of patients still develop metastasis after surgery.

Carbonic anhydrase IX (CAIX) is a newly discovered isoform of the carbonic anhydrase family, composed of acidic amino acids as a transmembrane glycoprotein. Located downstream of the VHL (von Hippel-Lindau) tumor suppressor gene, it is activated by the hypoxia-inducible factor-1 (HIF-1) pathway and plays a significant role in regulating cell proliferation and transformation. CAIX catalyzes the hydrolysis of carbon dioxide into bicarbonate and water, participating in acid-base balance regulation and modulating intracellular/extracellular pH. It is minimally expressed in normal tissues but highly expressed in hypoxic tumors such as RCC, promoting tumor growth and metastasis, and is closely associated with prognosis. Therefore, CAIX is a specific target for RCC, and its high tissue-specific expression holds critical importance for RCC diagnosis, staging, and treatment selection.

¹⁸F-NY104 is a novel PET imaging agent with a simple preparation process, whose yield and radiochemical purity meet clinical requirements. Preclinical studies demonstrate its specific binding to CAIX on tumor cell surfaces, superior pharmacokinetics and imaging performance compared to similar tracers, and promising potential for non-invasive, real-time, and comprehensive imaging diagnosis of CAIX-positive tumors. This project utilizes ¹⁸F-NY104 PET/CT to detect primary, recurrent, and metastatic RCC lesions, aiming to achieve comprehensive tumor localization and quantitative monitoring, thereby supporting early clinical diagnosis, staging, and restaging.

ELIGIBILITY:
Inclusion Criteria:

* (1)Capable of understanding and voluntarily signing the informed consent form; able to complete the trial in accordance with the protocol requirements; (2)Age 18-75 years; no gender restrictions; (3)Clinically diagnosed/suspected as renal cell carcinoma or clinically diagnosed/suspected recurrence/metastasis after RCC treatment; (4)At least 1 measurable solid lesion in the subject, which can be accurately and continuously measured using modified RECIST criteria (version 1.1); (5)ECOG performance status score of 0-2; (6)Laboratory parameters must meet:

  1. Hematology: WBC ≥4.0×10⁹/L or neutrophils ≥1.5×10⁹/L, PLT ≥100×10⁹/L, Hb ≥90g/L; PT or APTT ≤1.5×ULN (upper limit of normal);
  2. Liver and kidney function: T-Bil ≤1.5×ULN, ALT/AST ≤2.5×ULN or ≤5×ULN (for subjects with liver metastasis), ALP ≤2.5×ULN (if bone or liver metastasis present, ALP ≤4.5×ULN); BUN ≤1.5×ULN, SCr ≤1.5×ULN;
  3. Other routine tests within normal ranges or deemed acceptable by the investigator; (7)Expected survival ≥12 weeks; (8) Female subjects: Effective contraception (defined as sterilization, intrauterine hormone device, condoms, contraceptives/agents, abstinence, or partner vasectomy) must be used during the study and for 6 months post-study; Male subjects: Agreement to use contraception during the study and for 6 months post-study.

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study examination;
2. Patients with systemic or local severe infections or other serious comorbidities;
3. Severe hepatic or renal dysfunction;
4. Refusal to participate in this clinical study;
5. Patients with a history of allergy to any component of the imaging agent (including antibodies) or allergic constitution;
6. Childbearing-aged male or female subjects who cannot adopt effective contraception;
7. Women planning pregnancy, currently pregnant, or lactating;
8. Patients unable or unwilling to undergo PET/CT scanning;
9. Other subjects deemed ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort primarily included patients who were either clinically diagnosed with or suspected to have clear cell renal cell carcinoma (ccRCC), or those with suspected post-treatment recurrence or metastasis of ccRCC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No